CLINICAL TRIAL: NCT02317224
Title: Comparison of Safety and Efficacy Among "3-Hole" Subxiphorid Approach, Trans Sternal Approach and VATS in Surgical Treatment of Anterior Mediastinal Tumor
Brief Title: The Safety and Efficacy of "3-Hole" Subxiphorid Approach in the Treatment of Anterior Mediastinal Tumor
Acronym: 3-Hole
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Yongan Zhou, Associate Professor, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TangduH717544
Record Dates: First submitted 2014-11-26; First posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Thymectomy; Myasthenia Gravis
Keywords: 3-Hole approach; extended thymectomy; myasthenia gravis; safety; effectiveness
MeSH Terms: conditions — Myasthenia Gravis | interventions — Sternotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "3-Hole" subxiphorid and subcostal approach (Experimental): The patient were in the supine position with legs apart at about 45°, made a 2.0 cm incision below xiphoid process as the observation hole. Then made two 0.5cm operation holes along bilateral rib arch at midclavicular line, two trocars were inserted into the two holes under the guidance of B-ultrasound.After that, carbon dioxide was pumped into the anterior mediastinum, the pressure was maintained at 8 mmH2O, ultrasound scalpel and a grasping forceps were inserted through the operating ports respectively. Retrosternal space including bilateral lower poles of thymus, internal mammary arteries and phrenic nerves were exposed by both blunt and sharp dissection. Then ultrasound scalpel were used to separate the thymus and its surrounding fat tissue, cut off thymic veins by ultrasound scalpel.For patients with myasthenia gravis, bilateral mediastinal pleurae and the affected adipose tissues had been thoroughly removed.
  Interventions: Procedure: "3-Hole" subxiphorid and subcostal approach
- Trans sternal approach (Experimental)
  Interventions: Procedure: Trans sternal approach
- VATS approach (Experimental)
  Interventions: Procedure: VATS approach

INTERVENTIONS:
Procedure: "3-Hole" subxiphorid and subcostal approach — "3-Hole" subxiphorid and subcostal approach anterior mediastinum tumor resection
  Other Names: 3-Hole approach
  Arms: "3-Hole" subxiphorid and subcostal approach
Procedure: Trans sternal approach — Trans sternal approach anterior mediastinum tumor resection
  Other Names: median sternotomy
  Arms: Trans sternal approach
Procedure: VATS approach — Video-assisted thoracoscope anterior mediastinum tumor resection
  Other Names: Video-assisted thoracoscope
  Arms: VATS approach

SUMMARY:
Surgery plays an important role in the treatment of anterior mediastinum disease. The major surgical approaches include: cervical approach, mid-sternal approach, cervical combined mid-sternal approach and video-assisted thoracoscopic approach. The cervical approach is rarely adopted because of its restricted visual field. The cervical combined mid-sternal approach have a broader field of vision, given this advantage, the surgeon can remove the thymus and its surrounding fat tissue more thoroughly. But the trauma of this approach is much larger, and the postoperative complication is also a serious problem. The video-assisted thoracoscope is often adopted by left or right approach, this minimally invasive procedure can not remove anterior mediastinum fat thoroughly. In clinical practice, the investigators designed a new method named "3-Hole" subxiphoid approach. This study is designed to compare the safety and validity between this new method and others.

ELIGIBILITY:
Inclusion Criteria:

* MG with thymic hyperplasia, thymoma or other anterior mediastinum disease
* Masaoka stagingⅠ-Ⅱ
* Thymoma without MG
* Mass diameter <10cm
* Inform Consent Form is signed

Exclusion Criteria:

* Unable to tolerate surgery
* myasthenic crisis
* Masaoka staging Ⅲ-Ⅳ
* Patients who have undergone previous surgery or radiotherapy
* pregnancy , breastfeeding or younger than 18 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-08; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Amount of bleeding | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Measured by the difference between the wet weight and dry weight of surgical gauze
Rate of conversions to thoracotomy | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Only in "3-Hole" subxiphorid group and VATS group
Duration of operation | Participants will be followed for the duration of hospital stay, an expected average of 5 days
Mortality rate | up to 10 years
  Death caused by operation or complications
Overall survival | up to 10 years
  From randomization to any cause of death
Quality of life | up to 10 years after operation
  Measured by EORTC QLQ-C30 (version 3) scale
Number of Participants with Adverse Events | up to 8weekss afte operation

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu hospital, Xi'an, Shaanxi, China